CLINICAL TRIAL: NCT05200117
Title: Intra-observer Variability in the Assessment of Cervical Stiffness With the Pregnolia System
Brief Title: Pregnolia System Intra-observer Variability
Status: Completed | Type: Observational
Sponsor: Pregnolia AG (Industry)
Responsible Party: Sponsor
Other Study IDs: F-405-11 vs 3.0, 2023-07-21
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Cervix; Pregnancy; Cervical Stiffness
Keywords: Cervical Stiffness; Intra-Observer Variability; Pregnolia System; Cervical Stiffness Index; CSI; Stiffness measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nulliparous cohort: Cervical stiffness will be measured in the same subject sequentially between days and during the same day and at different gestational ages.
  Interventions: Device: Pregnolia System
- Multiparous cohort: Cervical stiffness will be measured in the same subject sequentially between days and during the same day and at different gestational ages.
  Interventions: Device: Pregnolia System

INTERVENTIONS:
Device: Pregnolia System — The cervical stiffness is measured with the Pregnolia System three times over a two-day period.

SUMMARY:
The Pregnolia System is a CE-marked medical device assessing the mechanical stiffness of cervical tissue in women. The Pregnolia Probe has been engineered to minimize the influence of differences in handling and technique by the user.

This project aims to study intra-observer variability of the Pregnolia System in pregnant women in the clinical setting.

Furthermore, a same day repeated measurement serves to investigate the time period needed to recover the pre-measurement stiffness state due to viscoelasticity of the cervical tissue.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Pregnant woman
* Singleton pregnancy
* 18 years or older
* Nulliparous cohort: nulliparous pregnant woman
* Multiparous cohort: multiparous pregnant woman

Exclusion Criteria:

* Lack of informed consent
* Placenta praevia totalis with haemorrhage (irrespective of severity)
* Severe vaginal bleeding
* Rupture of membranes before 34 weeks (to be excluded with pH test)
* Visible tissue scarring at 12 o'clock position on cervix
* Light bleeding (if the bleeding can be stopped, it is no longer an exclusion criterion)
* Cervical dilation ≥ 3 cm
* Cerclage or pessary in place

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women at gestational ages between 14+0 and 36+6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2023-12-17 (Actual)

PRIMARY OUTCOMES:
Cervical Stiffness Index | Measurements between 14+0 and 41+6 weeks gestational weeks
  Cervical Stiffness Index (CSI, in mbar) measured repeatedly after 2 to 4 hours and approximately 24 hours at three different locations on the uterine cervix.

SECONDARY OUTCOMES:
Cervical Stiffness Index (CSI, in mbar) | Measurements between 14+0 and 41+6 weeks gestational weeks
Elapsed time between | Measurements between 14+0 and 41+6 weeks gestational weeks
  The elapsed time between when the subject got out of bed until the measurements were taken
Device-related adverse events | Measurements between 14+0 and 41+6 weeks gestational weeks
  Device-related adverse events (incidence, severity, and seriousness)

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Frauenfeld, Frauenfeld, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided